CLINICAL TRIAL: NCT06289361
Title: Immunovirological Follow-up and Safety of HIV-infected Patients Receiving Lenacapavir Under Compassionate Access in France Between 01/01/2021 and 12/31/2023
Brief Title: Cohort IMEA 070 -Lenacapavir Compassional
Status: Active, not recruiting | Type: Observational
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Collaborators: Saint-Louis Hospital, Paris, France (Other); Bichat Hospital (Other); Saint Antoine University Hospital (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: IMEA 070
Record Dates: First submitted 2024-02-26; First posted 2024-03-01 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: HIV Infections
Keywords: Lenacapavir under compassionate access; France; Cohort
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Immunovirological follow-up and safety of HIV-infected patients receiving lenacapavir under compassionate access in France between 01/01/2021 and 12/31/2023

DETAILED DESCRIPTION:
Retrospective descriptive cohort of patients who received Lenacapavir under compassionate access in France with 50 patients in 25 sites in France

ELIGIBILITY:
Inclusion Criteria:

* Patients who received compassionate access to LEN between 01/01/2021 and 20/12/202

Exclusion Criteria:

* Absence of visits with virological assessment subsequent to inclusion visit
* Participant opposition to use of follow-up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already followed and identified in the centers and having received lenacapavir in compassionate access between January 01st, 2021 and December 20th, 2022
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
proportion of participants with plasma HIV RNA < 50 copies/ml 26 weeks after first LEN injection | Week 26

SECONDARY OUTCOMES:
incidence of side effects and laboratory abnormalities on LEN treatment | between week 26 and Week 52
evolution of HIV-1 or HIV-2 RNA over time | between week 26 and Week 52
evolution of CD4, CD8 lymphocyte counts and CD4/CD8 ratio over time | between week 26 and Week 52
Proportion of patients with capsid resistance mutations emergence at time of virological failure response) compared with initiation (D0) | between Week 26 and Week 52
Determination by multivariate analysis of factors associated with virological success 26 weeks after the first LEN injection factors associated with virological control 26 weeks after the first LEN injection | Week 26

CONTACTS AND LOCATIONS:
Locations (23):
- France (23):
  - Centre Hospitalier de la Côte Basque, Bayonne, France
  - Hôpital Béclère, Clamart, France
  - Hôpital de la Rochelle, La Rochelle, France
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, France
  - Hôpital Max Fourestier, Nanterre, France
  - CHU La Source, Orléans, France
  - Hôpital Félix Guyon, Saint-Denis, LA Reunion
  - Hopital Zobda Quitman, Fort-de-France, Martinique
  - Hopital Avicenne, Bobigny
  - Hôpital Pellegrin - Service de Médecine Interne et Maladies Infectieuses, Bordeaux
  - Hopital Saint-Andre, Bordeaux
  - Hopital Raymond Poincare, Garches
  - C.H.D de Vendee, La Roche-sur-Yon
  - André Mignot Hospital, Le Chesnay
  - Centre Hospitalier Bretagne Sud - Hôpital du Scorff, Lorient
  - CHU de Nice, Nice
  - Hôpital Hotel Dieu, Paris
  - Hopital Saint Antoine, Paris
  - Groupe Hospitalier Pitié-Salpêtrière - Service de Maladies Infectieuses et Tropicales, Paris
  - Hopital Necker, Paris
  - Bichat Hospital, Paris
  - Delafontaine, Saint-Denis
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No